CLINICAL TRIAL: NCT01211015
Title: Endoplasmic Reticulum (ER) Stress in Patients With Various Chronic Pulmonary Diseases
Brief Title: Endoplasmic Reticulum Stress in Chronic Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chonbuk National University (Other)
Responsible Party: Yong Chul Lee, Chonbuk National University Medical School
Other Study IDs: RCPD ER stress
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: ER Stress,; Chronic Airway Disorders,; Lung Cancer,; Interstitial Lung Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (2):
- Control group: healthy control group
- Disease group: asthma, COPD, ILD, lung malignancy

SUMMARY:
Aim: To investigate whether ER stress is implicated in the pathogenesis of various pulmonary disorders

Measurement:

1. Unfolded protein responses (UPRs) in blood (PBMCs)of patients

   1. CHOP
   2. GRP 78 and so on
2. Unfolded protein responses (UPRs) in blood (PBMCs)of healthy controls

   1. CHOP
   2. GRP 78 and so on

ELIGIBILITY:
Inclusion Criteria:

* > 18 yrs
* Definitive diagnosis as chronic pulmonary diseases by physician

Exclusion Criteria:

* Any other chronic medical illness such as DM, HTN, and other malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Control group
     * healthy control (volunteer)
  2. Disease group
     * chronic pulmonary lung diseases including asthma, COPD, ILD, and lung cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea